CLINICAL TRIAL: NCT06295796
Title: An Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics of MK-8527 in Participants With Moderate and Severe Renal Impairment
Brief Title: A Study of MK-8527 in Participants With Moderate and Severe Renal Impairment (MK-8527-008)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8527-008; MK-8527-008 (Other: MSD)
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Moderate Renal Impairment (Experimental): Participants with moderate renal impairment receive a single dose of MK-8527 on Day 1.
  Interventions: Drug: MK-8527
- Severe Renal Impairment (Experimental): Participants with severe renal impairment receive a single dose of MK-8527 on Day 1.
  Interventions: Drug: MK-8527
- Healthy (Experimental): Healthy participants receive a single dose of MK-8527 on Day 1.
  Interventions: Drug: MK-8527

INTERVENTIONS:
Drug: MK-8527 — Oral Capsule

SUMMARY:
The goal of this study is to evaluate the effect of moderate and severe renal impairment (RI) on the pharmacokinetics (PK), safety, and tolerability of MK-8527. There will be no hypothesis testing in the study.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

Moderate and Severe RI

* With the exception of RI, is in sufficient health for study participation.
* Has stable renal function.

Healthy

* Matches mean age to participants with moderate and severe RI.
* Has normal renal function.

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

All participants

* History of cancer (malignancy).
* Positive test results for Human-immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), or Hepatitis C virus (HCV).
* Had a major surgery or lost significant volume of blood within 56 days prior to dosing.
* Donated plasma within 7 days prior to dosing.

Moderate and Severe RI

* Failed renal transplant or had a nephrectomy.
* End stage renal disease requiring dialysis.
* Any significant arrhythmia or conduction abnormality.
* Has non-sustained or sustained ventricular tachycardia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Area under the concentration versus time curve from time 0 to last quantifiable sample (AUC0-last) of MK-8527 in plasma | Predose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 168 hours post dose
  AUC0-last of MK-8527 in plasma will be determined.
Area under the concentration versus time curve from time 0 to infinity (AUC0-inf) of MK-8527 in plasma | Predose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 168 hours post dose
  AUC0-inf of MK-8527 in plasma will be determined.
Maximum concentration (Cmax) of MK-8527 in plasma | Predose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 168 hours post dose
  Cmax of MK-8527 in plasma will be determined.
Time to Maximum concentration (Tmax) of MK-8527 in plasma | Predose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 168 hours post dose
  Tmax of MK-8527 in plasma will be determined.
Apparent terminal half-life (t1/2) of MK-8527 in plasma | Predose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 168 hours post dose
  t1/2 of MK-8527 in plasma will be determined.
Apparent Clearance (CL/F) of MK-8527 in plasma | Predose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 168 hours post dose
  CL/F of MK-8527 in plasma will be determined.
Apparent volume of distribution during terminal phase (Vz/F) of MK-8527 in plasma | Predose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 168 hours post dose
  Vz/F of MK-8527 in plasma will be determined.

SECONDARY OUTCOMES:
Number of participants who experience one or more adverse events (AEs) | Up to approximately 29 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants who discontinue study due to an AE | Up to approximately 29 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
AUC0-last of MK-8527-triphosphate (TP) in peripheral blood mononuclear cells (PBMCs) | Predose, 4, 12, 24, 48, 96, 120, 144, 168, 336, 504, 672 hours post dose
  AUC0-last of MK-8527-TP in PBMCs will be determined.
AUC0-inf of MK-8527-TP in PBMCs | Predose, 4, 12, 24, 48, 96, 120, 144, 168, 336, 504, 672 hours post dose
  AUC0-inf of MK-8527-TP in PBMCs will be determined.
Cmax of MK-8527-TP in PBMCs | Predose, 4, 12, 24, 48, 96, 120, 144, 168, 336, 504, 672 hours post dose
  Cmax of MK-8527-TP in PBMCs will be determined.
Concentration at 168 hours (C168) of MK-8527-TP in PBMCs | 168 hours post dose
  C168 of MK-8527-TP in PBMCs will be determined.
Concentration at 672 hours (C672) of MK-8527-TP in PBMCs | 672 hours post dose
  C672 of MK-8527-TP in PBMCs will be determined.
Tmax of MK-8527-TP in PBMCs | Predose, 4, 12, 24, 48, 96, 120, 144, 168, 336, 504, 672 hours post dose
  Tmax of MK-8527-TP in PBMCs will be determined.
t1/2 of MK-8527-TP in PBMCs | Predose, 4, 12, 24, 48, 96, 120, 144, 168, 336, 504, 672 hours post dose
  t1/2 of MK-8527-TP in PBMCs will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Research by Design ( Site 0001), Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com